CLINICAL TRIAL: NCT05273099
Title: Molecular Biomarkers Predicting Early Development of Endometrial Carcinoma: A Pilot Study
Brief Title: Molecular Biomarkers Predicting Early Development of Endometrial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Gennaro Scutiero, Principal Investigator, Università degli Studi di Ferrara
Other Study IDs: 170578
Record Dates: First submitted 2022-02-17; First posted 2022-03-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Cancer of Endometrium
Keywords: biomarkers; cancer gene mutations; endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Endometrium sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometrial carcinoma represents the most common gynaecological cancer and the sixth most frequent cancer among women worldwide. The 5-year survival of patients with stage I endometrial carcinoma is 75%-88% versus 50% for stage III or 15% for stage IV disease. Therefore, early detection could improve survival rates. Specifically, in the most prevalent, type 1 endometrial cancer develops from hyperplastic endometrium. The aim of the study was to evaluate the utility of cancer gene mutations from endometrial biopsies towards predicting synchronous or metachronous development of malignant lesions. The aim of the study was to evaluate whether endometrial biopsies could already carry mutations in cancer genes useful for predicting or anticipating subsequent cancer development

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* patients subjected to endometrial biopsies with previous histopathologically negative and subsequent histopathologically positive for endometrial carcinoma
* patient informed consent

Exclusion Criteria:

- Endometrial carcinoma patients without a previous non-tumour biopsy were excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with endometrial cancer and previous negative endometrial sample.
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mutation analyses on matched samples from female patients with a previous endometrial biopsy negative for cancer, followed by a subsequent biopsy positive for cancer | 1 year
  Mutation analyses performed on DNA isolated from formalin fixed, paraffin embedded samples retrieved for each patient by sequencing a panel of fifty genes (ABL1, AKT1, ALK, APC, ATM, BRAF, CDH1, CDKN2A, CSF1R, CTNNB1, EGFR, ERBB2, ERBB4, EZH2, FBXW7, FGFR1, FGFR2, FGFR3, FLT3, GNA11, GNAQ, GNAS, HNF1A, HRAS, IDH1, IDH2, JAK2, JAK3, KDR, KIT, KRAS, MET, MLH1, MPL, NOTCH1, NPM1, NRAS, PDGFRA, PIK3CA, PTEN, PTPN11, RB1, RET, SMAD4, SMARCB1, SMO, SRC, STK11, TP53, VHL) both on non-cancerous biopsies and on matched endometrial carcinoma biopsies.

SECONDARY OUTCOMES:
Integration of molecular results with clinico pathological data | 1 year
  Integration of molecular results with clinico pathological data

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Scutiero, MD, Principal Investigator — Department of Morphology, Surgery and Experimental Medicine, University of Ferrara, Ferrara, Italy
Locations (1):
- Section of Obstetrics and Gynecology, Department of Morphology, Surgery and Experimental Medicine, University of Ferrara, Ferrara, Italy, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakkum-Gamez JN, Wentzensen N, Maurer MJ, Hawthorne KM, Voss JS, Kroneman TN, Famuyide AO, Clayton AC, Halling KC, Kerr SE, Cliby WA, Dowdy SC, Kipp BR, Mariani A, Oberg AL, Podratz KC, Shridhar V, Sherman ME. Detection of endometrial cancer via molecular analysis of DNA collected with vaginal tampons. Gynecol Oncol. 2015 Apr;137(1):14-22. doi: 10.1016/j.ygyno.2015.01.552. Epub 2015 Feb 10. PMID 25677060
- [Background] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Suhaimi SS, Ab Mutalib NS, Jamal R. Understanding Molecular Landscape of Endometrial Cancer through Next Generation Sequencing: What We Have Learned so Far? Front Pharmacol. 2016 Nov 1;7:409. doi: 10.3389/fphar.2016.00409. eCollection 2016. PMID 27847479